CLINICAL TRIAL: NCT02484131
Title: Bone Health Management for Women Diagnosed With Breast Cancer: A Pilot Study
Brief Title: Bone Health Management for Women Diagnosed With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Olivia Tseng, MD, MD. MSc, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H15-00849
Record Dates: First submitted 2015-06-12; First posted 2015-06-29 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Osteoporosis; Breast Cancer
Keywords: Osteoporosis; DXA Screening; Women; Breast Cancer; Survivors; Educational materials; Personal choices on delivery methods
MeSH Terms: conditions — Osteoporosis; Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: data analyst
Oversight: Data Monitoring Committee: No

ARMS (3):
- Educational materials/mail (Experimental): Participants in this group will receive educational materials by mail on the first day of the follow-up period.
  Interventions: Behavioral: Educational materials/mail
- Educational materials/participant choice (Experimental): Participants in this group will receive educational materials by participant choice on the first day of the follow-up period.
  Interventions: Behavioral: Educational materials/participant choice
- Control (No Intervention): Participants in this group will not receive any educational materials during hte follow-up period. Educational materials will be sent by mail after the completion of this study.

INTERVENTIONS:
Behavioral: Educational materials/mail — Participants in this group will receive any educational materials by mail during hte follow-up period.
  Arms: Educational materials/mail
Behavioral: Educational materials/participant choice — Participants in this group will not receive any educational materials by participant choice during hte follow-up period.
  Arms: Educational materials/participant choice

SUMMARY:
The purpose of this study is to test the feasibility of the study protocol. The study protocol was designed to evaluate questions - "Do educational materials improve dual x-ray absorptiometry (DXA) screening rates for women diagnosed with breast cancer" and "Does educational materials delivered by the participant's selected choice change DXA screening rates compared to the conventional mail method?".

DETAILED DESCRIPTION:
"Bone health management" for osteoporosis is important for women diagnosed with breast cancer. Osteoporosis can lead to bones breaking easily. Broken bones may make living independently challenging. Effective bone health management can reduce the risk of broken bones. This study will examine whether providing "osteoporosis information" to women diagnosed with breast cancer will promote their bone health management. With the current advance in technology, people are more interested in receiving information by email or smartphone text messaging. This study will also examine whether delivering osteoporosis information in different ways will change bone health management.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Is 65-75 year old on July 1st, 2015
* Lives in British Columbia (BC), Canada
* Reads and understands the information provided in English
* Was diagnosed with breast cancer prior to July 1st, 2012
* Is not receiving surgery, radiation or chemotherapy for any cancers
* Has not had breast cancer spread beyond her breast(s) and nearby lymph nodes
* Has not had screening tests after July 1st, 2012
* Is not taking medications prescribed by doctors for osteoporosis

Exclusion criteria:

* Is medically unfit for preventive care (death, cognitive impairment, nursing home admission, severe mental illness, etc), which will be determined by their family doctors
* Have terminated patient-doctor relationship with her family doctor who is indicated in our record

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
DXA screening rates | 6 months

SECONDARY OUTCOMES:
Percentage of participants diagnosed with osteoporosis | 6 months
Percentage of participants initiating osteoporosis medication | 6 months
Changes in Calcium in take | 6 months
  measured as mg per week using validated questionnaires
Changes in vitamin D status | 6 months
  measured as scores using validated questionnaires
Changes in exercise patterns | 6 months
  measured as scores using validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dawes, MD, PhD, Principal Investigator — University of British Columbia; John J. Spinelli, PhD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided